CLINICAL TRIAL: NCT06601153
Title: Health Improvements by Understanding Residual Risk in CAd and NEw Targets for Prevention/treatment - HURRICANE
Brief Title: Health Improvements by Understanding the Determinants of Residual Risk in Coronary Artery Disease and New Targets for Prevention and Treatment
Acronym: HURRICANE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Toscana Gabriele Monasterio (Other)
Collaborators: CNR Institute of Clinical Physiology, Pisa, Italy (Unknown); IRCCS SYNLAB SDN, Naples, Italy (Unknown)
Responsible Party: Principal Investigator, Danilo Neglia, MD, PhD, Fondazione Toscana Gabriele Monasterio
Other Study IDs: PNRR-MAD-2022-12376550
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: coronary artery disease (CAD); cardiac CT (CCT); cardiovascular risk factors; atherogenic dyslipidemia; insulin resistance (IR); molecular medicine; genetics.
MeSH Terms: conditions — Coronary Artery Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma, serum and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort of 561 patients with suspected CAD: All patients with suspected CAD with available blood samples stored in bio-banks and interpretable CCT stored in imaging repositories.
  Interventions: Diagnostic Test: Cardiac CT
- Prospective cohort od 400 patients with suspected CAD: All patients with suspected CAD in whom with blood samples will be collected and stored in bio-banks and CCT will be acquired and stored in imaging repositories.
  Interventions: Diagnostic Test: Cardiac CT

INTERVENTIONS:
Diagnostic Test: Cardiac CT — Cardiac CT to characterize coronary atherosclerosis
  Other Names: Computed Tomography Coronary Angiography

SUMMARY:
Current medical treatments, in patients with stable coronary artery disease (CAD), mainly target established risk factors and are able to reduce morbidity and mortality but still leave a substantial residual risk of coronary artery disease progression and events. The main hypothesis of this study is that metabolic derangement, including pre-diabetes, elevated levels of triglycerides, low levels and functionality of high-density lipoprotein cholesterol, often associated with a chronic inflammatory state, is a currently unrecognized and undertreated conditon which could be the most relevant determinant of residual risk.

The goal of HURRICANE observational study is to discover specific individual genetic/molecular profiles subtending emerging cardiometabolic and vascular risk patterns and associating with a more severe and progressive coronary artery disease. We will thus develop and preliminary validate new predictive models for the recognition of high-risk patients and explore possible new targets for individualized preventive treatment.

The severity, extent and progression of coronary plaques will be assessed by qualitative and quantitative analysis of cardiac computed tomography (CCT) performed in retrospective and prospective cohorts of patients with stable coronary disease.

DETAILED DESCRIPTION:
HURRICANE is an observational clinical study, performed in retrospective and prospective cohorts of patients with stable CAD, to assess the role of emerging cardiometabolic and vascular risk determinants to predict severe and progressive coronary atherosclerosis documented by advanced CCT imaging.

The population of the retrospective study consists of two parallel, independent groups of patients enrolled in previous clinical trials focused on blood and CCT biomarkers of CAD. All participants are assessed for eligibility to the current study which includes in particular availability of blood samples in bio-bank and of interpretable CCT exams. For each cohort and for the whole retrospective population (561 patients) clinical variables (demographic data, cardiovascular risk factors, history of previous CAD, symptoms and medications) and conventional circulating biomarkers (lipid and glucose metabolism, systemic inflammation, liver and kidney function) are recorded. The coronary imaging variables which will provide the disease presence and severity end-points will be derived from qualitative and semiquantitative analyses of CCT exams according to CAD-RADS 2.0 classification system.

The population of the prospective longitudinal study will include 400 patients referred at IRCCS SYNLAB SDN in Naples and FTGM in Pisa, over a 12 months period, to a clinically indicated CCT for suspected CAD, signing a written informed consent and fulfilling Inclusion and exclusion criteria. At baseline, patients will be characterized as in the retrospective study (same clinical variables, conventional circulating biomarkers and CCT imaging variables) and blood samples will be collected and stored in the dedicated Bio-Bank for advanced genetic/molecular analyses. They will be submitted to monitoring visits and a last follow-up visit at 12 months when compliance to medical treatment and events will be registered. A second blood sample will be collected and stored in dedicated Bio-Bank for advanced molecular analyses. A second CCT scan will be performed at 12 months with the same scanner, at the same institution, by the use of a state-of-the art CCT technology with high spatial and temporal resolution to provide quantitative measurements of coronary plaque volumes and coronary plaque composition which will be used to define the disease progression end-points.

Qualitative and semiquantitative analyses of CCT exams will be performed by radiologists according to CAD-RADS 2.0 classification systemin both the retrospective and prospective populations. In the prospective population, CCT images at enrollment and follow-up will also be quantitatively analyzed to define evolving CAD phenotypes. Quantitative analysis will be performed on visually identified plaques using a dedicated software package (QAngio CT Research Edition version 3.1.2.0, Medis Medical Imaging Systems, Leiden, the Netherlands) to generate detailed output on the lumen and plaque statistics, including the degree of stenosis, lesion length, vessel volume, plaque burden, plaque volume, and plaque components (according to the virtual histology classification: dense calcium, necrotic core, fibrous-fatty, fibrous, and media). Additional CT-derived parameters will also be assessed, in particular epicardial and perivascular adipose tissue, to be tested in the predictive models of CAD evolution and to be entered in a Machine Learning data analysis as potential variables of the pathophysiologic CAD network.

Circulating biomarkers will be evaluated by standard methodologies of clinical chemistry laboratories at the two participant clinical centers and specific circulating biomarkers will be analyzed at the IFC-CNR Core-Lab in both the retrospective and the prospective populations. In particular, additional markers of lipid metabolism and adipose tissue function, endothelial function and atherosclerotic burden will be evaluated by dedicated immunoassays, while markers of myocardial damage/function will be evaluated by automatized immunoassays. The inflammatory profile will be assessed by multiplex cytokine screens."Omics" analyses, in both populations, will include lipidomic, with the assessment of circulating lipid species using mass spectrometry, and genetic profiling by GWAS (Genome-Wide Association Study) performed by an external provider (Genomix4Life) using new generation microarray technology to genotype single-nucleotide variants (SNVs). In representative extreme groups of patients from the prospective population, a specific panel of 88 candidate genes involved in lipid/glucose homeostasis, endothelial/vascular function and systemic inflammation, together with other relevant genes emerging from the GWAS analysis, will be sequenced for known and unknown variants at FTGM by NGS (Next Generation Sequencing) approach. The library preparation for NGS will be performed using the Illumina DNA Prep with Enrichment Kit. Base-Space Variant Interpreter software will be used to annotate, filter and interpret the variants. The degree of pathogenicity will be also assessed on VarSome (https://varsome.com) and GWAS Catalog (https://www.ebi.ac.uk/gwas/), search engines and impact analysis tools for human genetic variation. The variants identified as pathogenetically relevant, in the subjects with extreme phenotypes will then be assessed in the rest of the population. Moreover, miRNAs, putatively associated with relevant gene variants and screened by in silico bioinformatic analysis, will be assessed by qPCR.

ELIGIBILITY:
RETROSPECTIVE STUDY

Inclusion Criteria:

* patients with known or suspected stable CAD who underwent CCT for the registered studies "SMARTool" or "Studio di biomarcatori in vivo ed in vitro"
* fully accessible CCT image files and whole blood and plasma/serum aliquots stored in BioBank
* written informed consent

Exclusion Criteria:

* overt heart failure (NYHA Class III-IV) and/or reduced systolic LV function (LVEF<40%)
* relevant comorbid conditions limiting expected survival to less than 1 year
* CCT exam of suboptimal quality

PROSPECTIVE STUDY

Inclusion Criteria:

* patients with suspected stable CAD clinically referred for a first diagnostic CCT
* fully accessible CCT image files and whole blood and plasma/serum aliquots stored in BioBank
* written informed consent

Exclusion Criteria:

* history of previous CAD or major cardiovascular events
* overt heart failure (NYHA Class III-IV) and/or reduced systolic LV function (LVEF<40%)
* relevant comorbid conditions limiting expected survival to less than 1 year
* CCT exam of suboptimal quality

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RETROSPECTIVE STUDY From the 684 patients with suspected or known stable CAD, referred to IRCCS SYNLAB SDN in Naples between July 2018 and March 2022 for clinically indicated CCT and enrolled in a previous study (Observational Study 7/18 OSS SDN), 376 patients meeting all eligibility criteria are included in the HURRICANE retrospective study population.
  From the 263 patients with suspected or known stable CAD, undergoing CCT at FTGM in Pisa from September 2012 to October 2913 and enrolled in a previous study (SMARTool, HORIZON 2020-689068), 185 patients meeting all eligibility criteria complete the HURRICANE retrospective study population.
  PROSPECTIVE STUDY The population of the prospective longitudinal study will include 400 patients referred at IRCCS SYNLAB SDN in Naples and FTGM in Pisa, over a 12 months period, to a clinically indicated CCT for suspected CAD, meeting all eligibility criteria and signing a written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 961 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | In the prospective Study patients will be evaluated at baseline and follow-up within a18 months time frame.
  The primary objective is the development (retrospective study) and validation (prospective study) of new integrated clinical and molecular/genetic predictive models of severity and extent of CAD defined by CCT in patients with stable disease. Developed models will be extended (prospective study) to the prediction of progression (at 1-year follow-up) of CAD phenotypes occurring despite OMT. The hypothesis is that these models, including specific molecular markers (assessed by traditional laboratory as well as by "omics" approaches) of emerging cardiometabolic and vascular risk, could predict CAD severity/extent and progression more accurately than other traditional risk models.

SECONDARY OUTCOMES:
Secondary Objective | In the prospective Study selected groups of patients will be evaluated at baseline and follow-up within a18 months time frame.
  The secondary objective is to perform a pathophysiologic sub study in selected groups of patients, from the prospective population, with extreme cardiometabolic and coronary disease phenotypes. The hypothesis is that a specific characterization, focused on relevant molecules and genes involved in lipid/glucose homeostasis, endothelial/vascular function and chronic low-grade systemic inflammation, in selected groups of patients with/without clinically defined patterns of high cardiometabolic/vascular risk and with/without CCT defined phenotypes of high CAD risk may unveil pathophysiological associations yet unrecognized because diluted by multiple other confounding variables in the modelling approach performed in non-selected populations.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Neglia, MD, PhD, Study Chair — Fondazione Toscana Gabriele Monasterio
Locations (2):
- Italy (2):
  - Fondazione Toscana Gabriele Monasterio, Pisa, Italy
  - Irccs Synlab Sdn, Napoli

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing will be evaluated and decided together with the Institutions involved and in agreement with the rules of the competent Ethics Committees and of Italian Ministry of Health for PNRR funded prjects

REFERENCES:
- [Background] Cademartiri F, Meloni A, Pistoia L, Degiorgi G, Clemente A, Gori C, Positano V, Celi S, Berti S, Emdin M, Panetta D, Menichetti L, Punzo B, Cavaliere C, Bossone E, Saba L, Cau R, Grutta L, Maffei E. Dual-Source Photon-Counting Computed Tomography-Part I: Clinical Overview of Cardiac CT and Coronary CT Angiography Applications. J Clin Med. 2023 May 23;12(11):3627. doi: 10.3390/jcm12113627. PMID 37297822
- [Background] Neglia D, Liga R, Gimelli A, Podlesnikar T, Cvijic M, Pontone G, Miglioranza MH, Guaricci AI, Seitun S, Clemente A, Sumin A, Vitola J, Saraste A, Paunonen C, Sia CH, Paleev F, Sade LE, Zamorano JL, Maroz-Vadalazhskaya N, Anagnostopoulos C, Macedo F, Knuuti J, Edvardsen T, Cosyns B, Petersen SE, Magne J, Laroche C, Berle C, Popescu BA, Delgado V; EURECA Investigators. Use of cardiac imaging in chronic coronary syndromes: the EURECA Imaging registry. Eur Heart J. 2023 Jan 7;44(2):142-158. doi: 10.1093/eurheartj/ehac640. PMID 36452988
- [Background] Neglia D, Caselli C, Maffei E, Cademartiri F, Meloni A, Bossone E, Saba L, Lee SE, Sung JM, Andreini D, Al-Mallah MH, Budoff MJ, Chinnaiyan K, Choi JH, Chun EJ, Conte E, Gottlieb I, Hadamitzky M, Kim YJ, Lee BK, Leipsic JA, Marques H, de Araujo Goncalves P, Pontone G, Shin S, Stone PH, Samady H, Virmani R, Narula J, Shaw LJ, Bax JJ, Lin FY, Min JK, Chang HJ. Rapid Plaque Progression Is Independently Associated With Hyperglycemia and Low HDL Cholesterol in Patients With Stable Coronary Artery Disease: A PARADIGM Study. Circ Cardiovasc Imaging. 2024 Jul;17(7):e016481. doi: 10.1161/CIRCIMAGING.123.016481. Epub 2024 Jul 16. PMID 39012946
- [Background] Caselli C, De Caterina R, Smit JM, Campolo J, El Mahdiui M, Ragusa R, Clemente A, Sampietro T, Clerico A, Liga R, Pelosi G, Rocchiccioli S, Parodi O, Scholte A, Knuuti J, Neglia D; EVINCI and SMARTool. Triglycerides and low HDL cholesterol predict coronary heart disease risk in patients with stable angina. Sci Rep. 2021 Oct 20;11(1):20714. doi: 10.1038/s41598-021-00020-3. PMID 34671067
- [Background] Neglia D, Aimo A, Lorenzoni V, Caselli C, Gimelli A. Triglyceride-glucose index predicts outcome in patients with chronic coronary syndrome independently of other risk factors and myocardial ischaemia. Eur Heart J Open. 2021 Jul 24;1(1):oeab004. doi: 10.1093/ehjopen/oeab004. eCollection 2021 Aug. PMID 35919094
- [Background] Di Giorgi N, Michelucci E, Smit JM, Scholte AJHA, El Mahdiui M, Knuuti J, Buechel RR, Teresinska A, Pizzi MN, Roque A, Poddighe R, Parodi O, Pelosi G, Caselli C, Neglia D, Rocchiccioli S. A specific plasma lipid signature associated with high triglycerides and low HDL cholesterol identifies residual CAD risk in patients with chronic coronary syndrome. Atherosclerosis. 2021 Dec;339:1-11. doi: 10.1016/j.atherosclerosis.2021.11.013. Epub 2021 Nov 11. PMID 34801858
- [Derived] Caselli C, Occhipinti M, Pane K, De Gori C, Rocchiccioli S, Botto N, Prontera C, Cavaliere C, Ragusa R, Vecoli C, Sansone F, Passaro E, Ceccherini E, Morlando A, Clemente A, Franzese M, Maffei E, Punzo B, Gimelli A, Cademartiri F, Neglia D. Health improvements by understanding residual risk in coronary artery disease and new targets for prevention/treatment: rationale and research protocol of the HURRICANE project. Eur Heart J Open. 2025 Jan 28;5(1):oeaf005. doi: 10.1093/ehjopen/oeaf005. eCollection 2025 Jan. PMID 39949422